CLINICAL TRIAL: NCT03602378
Title: Quality of Life and Stress in Parents of Children With Developmental Disabilities and Chronic Disease
Brief Title: QoL and Stress in Parents of Children With Developmental Disabilities and Chronic Disease
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Split, School of Medicine (Other)
Collaborators: General Hospital Zadar (Other)
Responsible Party: Principal Investigator, Ivana Kolcic, MD, PhD, Associate Professor in Epidemiology Centre for Global Health & Department of Public Health Medical School, University of Split, University of Split, School of Medicine
Other Study IDs: 2181-198-03-04-18-0014
Record Dates: First submitted 2018-06-04; First posted 2018-07-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Developmental Disability; Chronic Disease; Down Syndrome; Autism Spectrum Disorder; Pervasive Developmental Disorder; Cerebral Palsy; Diabetes Mellitus, Type 1; Epilepsy; Asthma; Stress
Keywords: Parents; Quality of life; Stress; Children with developmental disability; Children with chronic disease; Cortisol; Heart rate variability; Advanced glycation end products; Sleep quality; Family cohesion; Stigma; Resilience; Anxiety; Depression; Self Esteem
MeSH Terms: conditions — Developmental Disabilities; Chronic Disease; Down Syndrome; Autism Spectrum Disorder; Child Development Disorders, Pervasive; Cerebral Palsy; Diabetes Mellitus, Type 1; Epilepsy; Asthma; Sleep Initiation and Maintenance Disorders; Social Stigma; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parents of children with disability: parents of children with developmental disabilities (Down syndrome, autism spectrum disorder, pervasive developmental disorder, cerebral palsy), age 20-50, salivary cortisol, Holter Medilog AR12 Plus, Polar V800, AGE reader
  Interventions: Diagnostic Test: salivary cortisol; Device: Holter Medilog AR12 Plus; Device: Polar V800; Device: AGE reader
- Parents of children with chronic disease: parents of children chronic disease (diabetes mellitus type 1, epilepsy, asthma), age 20-50, salivary cortisol, Holter Medilog AR12 Plus, Polar V800, AGE reader
  Interventions: Diagnostic Test: salivary cortisol; Device: Holter Medilog AR12 Plus; Device: Polar V800; Device: AGE reader
- Parents of healthy children: parents of healthy children, age 20-50, salivary cortisol, Holter Medilog AR12 Plus, Polar V800, AGE reader
  Interventions: Diagnostic Test: salivary cortisol; Device: Holter Medilog AR12 Plus; Device: Polar V800; Device: AGE reader

INTERVENTIONS:
Diagnostic Test: salivary cortisol — 5 samples of saliva (first sample before around 22:00 and other samples the next morning, after awakening (00, 15, 30 and 60 minutes).
Device: Holter Medilog AR12 Plus — Holter Medilog AR12 Plus - electrocardiogram during 5 minutes for measuring HRV
Device: Polar V800 — Polar V800 with sensor - during 5 minutes for measuring HRV
  Other Names: Polar V800 with sensor
Device: AGE reader — for measuring Advanced Glycation End products (AGEs)
  Other Names: Advanced glycation end products reader; AGEs reader

SUMMARY:
The aim of this cross-sectional study is to investigate the level of stress and quality of life in parents of children with developmental disabilities (Down syndrome, autism spectrum disorder, pervasive developmental disorder, cerebral palsy) and parents of children chronic diseases (diabetes mellitus type 1, epilepsy, asthma) compared to parents of healthy children.

The investigators will analyze the level of stress, quality of life, self-esteem, optimism, resilience, happiness, stigmatization, depression, anxiety, sleep quality, parenting challenges and some physiological indicators of the stress such as level of cortisol and heart rate variability. Also, the investigators will measure Advanced Glycation End products (AGEs) in the skin.

The investigators assume that parents of children with developmental disabilities and chronic diseases have higher level of stress and lower quality of life compared to the parents of healthy children.

DETAILED DESCRIPTION:
Participants will be parents of children with a pervasive developmental disorder (autistic spectrum disorder), Down syndrome, cerebral palsy, epilepsy, diabetes mellitus type 1, asthma, and parents of healthy children (without difficulty and chronic disease - control group).

The investigators will examine the level of stress and quality of life in parents of children with developmental and chronic illnesses, compared to parents of healthy children, adjusting for the effect of confounding factors.

Data collection will be conducted using the questionnaire to assess personal quality of life, family quality of life, general and parental stress levels. Additionally, potential confounding or mediating factors will be measured and taken into account: stress resilience, cohesion, self-esteem, optimism, perception of happiness, stigmatization, depression, anxiety, sleep quality and parenting challenges. Also, socio-demographics parameters, short medical history, lifestyle habits and the perception of life difficulties will be assessed. The questionnaire will be filled by paper-pencil method with anticipated duration of about 45 minutes.

The investigators will also measure several physiological indicators - salivary cortisol, heart rate variability, blood pressure and Advanced Glycation End products (AGEs).

Saliva will be taken in order to analyze the cortisol level, using Salivette Sarstedt REF 51.1534.500. Participants will be taken five saliva samples during the day because of the physiological variability of cortisol (first one around 22:00 hours, second right after waking up, then 15, 30 and 60 minutes after awaking). Each subject will receive detailed instructions on how to take saliva, with written instructions. Thirty minutes before sampling, the subjects has to restrain from eating, drinking, smoking or brushing teeth. In case of acute illness, inflammation or disease in the oral cavity, the sampling will be delayed. After taking the sample, tubes will be stored in the refrigerator. In the laboratory, the sample will be centrifuged for two minutes to remove saliva from cotton, and saliva samples will be frozen. Cortisol analysis will be done using ECLIA (Electrochemiluminous Absorption Method).

The electrocardiogram (ECG) will be recorded using the Medilog AR12 Plus Holter device, which will also be used to record heart rate variability (HRV) during 5 minutes. HRV will also be recorded using the Polar V800 (also during 5 minutes). Kubios software will be used for HRV analysis.

AGE Reader, a non-invasive device will be used for measuring the autofluorescence in the skin, reflecting the level of Advanced Glycation End products (AGEs).

Omrom M6 Comfort is an automatic device which will be used to measure blood pressure and pulse.

Anthropometric parameters will be measured (body weight, height, neck circumference, waist and hip circumference).

Statistical analysis will be carried out using statistical program MedCalc. Initial analysis of results will include analysis of the distribution of variables using the Kolmogorov-Smirnov test. If the distribution of numerical variables will be normal, parametric statistics will be applied. The confounding factors will be controlled by using appropriate statistical tests.

Participation of parents in this study is voluntary. If a parent decides to participate in this study, the code will be assigned. In that way, all data, measured parameters, and saliva samples will be encoded, and the personal data of the respondents will be completely invisible. It will not be possible to identity an individual parent. All researchers must and will be protecting confidentiality of data.

ELIGIBILITY:
Inclusion Criteria:

* subject are parents between 20 and 50 years,
* subject are parents of the child with developmental disability (Down syndrome, autism spectrum disorder, pervasive developmental disorder, cerebral palsy) or chronic disease (diabetes mellitus type 1, epilepsy, asthma) - the ages of the child between 4 and 12 years.

Exclusion Criteria:

* severe psychiatry and severe chronic illnesses of parents
* ischemic heart disease
* cardiomyopathy
* heart arrhythmia
* malignant hypertension
* diabetic neuropathy
* transplantation of heart and other organs
* tetraplegia
* diseases of the hypothalamus and pituitary and adrenal gland
* corticosteroid therapy
* antiarrhythmic therapy
* therapy of β-blockers
* therapy of sedatives
* therapy of anxiolytics
* chemotherapy
* night shift work
* breastfeeding (active or completed within less 6 months)
* pregnancy
* diagnose of child less than 6 months
* parents of children with other severe chronic or rare diseases such as malignant disease, haemophilia, phenylketonuria, neurofibromatosis.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Parents of children with Down syndrome, pervasive developmental disorder (autistic spectrum disorder), cerebral palsy, epilepsy, diabetes type 1, asthma, and parents of healthy children (without difficulties and chronic diseases - control group).
Sampling Method: Probability Sample
Enrollment: 592 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-04-02 (Estimated); Study Completion 2021-05-02 (Estimated)

PRIMARY OUTCOMES:
Quality of life in parents of children with developmental disability and chronic disease, and healthy children. | 1 day
  Subjects will complete the questionnaires about quality of life. A total 26 item in the WHOQOL-BREF produces four domain scores: physical, psychological, social relationships and environment domain (Likert type scale ranging from 1- strongly disagree to 5 - strongly agree).
Stress in parents of children with developmental disability and chronic disease, and healthy children. | 1 days
  Subjects will complete the questionnaires about parental stress. Parental Stress Scale consists of 18 item self report scale (Likert type scale ranging from 1-strongly disagree, 2-disagree, 3-undecided, 4-agree 5-strongly agree). Items represent positive (e.g. emotional benefits, personal development) and negative (demands on resources, restrictions) themes of parenthood.

SECONDARY OUTCOMES:
Family quality of life | 1 day
  A total 25 items in FQOL scale keyed for five domains scores: family interaction, parenting, emotional well-being, physical / material well-being and disability-related support (Likert type scale satisfaction are rated on a 5-point scale, where 1- very dissatisfied, 3-neither satisfied nor dissatisfied, and 5-very satisfied). Scores are scaled in a positive direction (i.e. higher scores denote higher quality of life).
Perceived Stress Scale | 1 day
  Perceived Stress Scale consists of 10 items (Likert type scale ranging from 0-never, 1-almost never, 2-sometimes,3-fairly often, 4-very often). Higher scores indicating greater levels of stress.
Salivary cortisol concentration in parents of children with developmental disability, chronic disease and parents of healthy children. | 1 day
  5 samples of saliva (first sample before around 22:00 and other samples the next morning, after awakening (00, 15, 30 and 60 minutes)).
Heart rate variability in parents of children with developmental disability, chronic disease and parents of healthy children | 1 day
  Holter Medilog AR12 Plus - electrocardiogram and Polar V800 with sensor - during 5 minutes
Advanced glycation end products in parents of children with developmental disability, chronic disease and parents of healthy children. | 1 day
  AGE reader for measuring advanced glycation end products. Higher results indicating greater cardiovascular risk.

CONTACTS AND LOCATIONS:
Overall Officials: MARIJA LJUBICIC, RN, MSN, Principal Investigator — General hospital Zadar, Department of Pediatrics; IVANA KOLCIC, MD, PhD, Principal Investigator — University of Split, School of Medicine
Locations (2):
- Croatia (2):
  - University Hospital Split, Split
  - Ivana Kolcic, Split

IPD SHARING:
Plan to Share IPD: Undecided
Identified participants for outcome measures

REFERENCES:
- [Background] Kleinman JM, Robins DL, Ventola PE, Pandey J, Boorstein HC, Esser EL, Wilson LB, Rosenthal MA, Sutera S, Verbalis AD, Barton M, Hodgson S, Green J, Dumont-Mathieu T, Volkmar F, Chawarska K, Klin A, Fein D. The modified checklist for autism in toddlers: a follow-up study investigating the early detection of autism spectrum disorders. J Autism Dev Disord. 2008 May;38(5):827-39. doi: 10.1007/s10803-007-0450-9. PMID 17882539
- [Background] Turner LM, Stone WL. Variability in outcome for children with an ASD diagnosis at age 2. J Child Psychol Psychiatry. 2007 Aug;48(8):793-802. doi: 10.1111/j.1469-7610.2007.01744.x. PMID 17683451
- [Background] Eaves LC, Ho HH. The very early identification of autism: outcome to age 4 1/2-5. J Autism Dev Disord. 2004 Aug;34(4):367-78. doi: 10.1023/b:jadd.0000037414.33270.a8. PMID 15449513
- [Background] Bella GP, Garcia MC, Spadari-Bratfisch RC. Salivary cortisol, stress, and health in primary caregivers (mothers) of children with cerebral palsy. Psychoneuroendocrinology. 2011 Jul;36(6):834-42. doi: 10.1016/j.psyneuen.2010.11.005. Epub 2010 Dec 10. PMID 21146316
- [Background] Stalder T, Kirschbaum C, Kudielka BM, Adam EK, Pruessner JC, Wust S, Dockray S, Smyth N, Evans P, Hellhammer DH, Miller R, Wetherell MA, Lupien SJ, Clow A. Assessment of the cortisol awakening response: Expert consensus guidelines. Psychoneuroendocrinology. 2016 Jan;63:414-32. doi: 10.1016/j.psyneuen.2015.10.010. Epub 2015 Oct 20. PMID 26563991
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Billman GE. Heart rate variability - a historical perspective. Front Physiol. 2011 Nov 29;2:86. doi: 10.3389/fphys.2011.00086. eCollection 2011. PMID 22144961
- [Background] Baba M, Ohkura M, Koga K, Nishiuchi K, Herrera LR, Matsuse R, Inoue T. Analysis of salivary cortisol levels to determine the association between depression level and differences in circadian rhythms of shift-working nurses. J Occup Health. 2015;57(3):237-44. doi: 10.1539/joh.14-0079-OA. Epub 2015 Mar 6. PMID 25752657
- [Background] Karhula K, Harma M, Sallinen M, Lindholm H, Hirvonen A, Elovainio M, Kivimaki M, Vahtera J, Puttonen S. Salivary cortisol and alpha-amylase: Is there consistency between psychosocial stress test and burdensome work shifts? J Occup Environ Hyg. 2017 Dec;14(12):1003-1010. doi: 10.1080/15459624.2017.1350786. PMID 28692340
- [Background] Niu SF, Chung MH, Chu H, Tsai JC, Lin CC, Liao YM, Ou KL, O'Brien AP, Chou KR. Differences in cortisol profiles and circadian adjustment time between nurses working night shifts and regular day shifts: A prospective longitudinal study. Int J Nurs Stud. 2015 Jul;52(7):1193-201. doi: 10.1016/j.ijnurstu.2015.04.001. Epub 2015 Apr 8. PMID 25900684
- [Background] Simon CD, Adam EK, McKinney CO, Krohn JB, Shalowitz MU. Breastfeeding, Bed-Sharing, and Maternal Cortisol. Clin Pediatr (Phila). 2016 May;55(5):470-8. doi: 10.1177/0009922815601981. Epub 2015 Sep 1. PMID 26330120
- [Background] Tu MT, Lupien SJ, Walker CD. Diurnal salivary cortisol levels in postpartum mothers as a function of infant feeding choice and parity. Psychoneuroendocrinology. 2006 Aug;31(7):812-24. doi: 10.1016/j.psyneuen.2006.03.006. Epub 2006 May 23. PMID 16716531
- [Background] Rogers SL, Hughes BA, Tomlinson JW, Blissett J. Cortisol metabolism, postnatal depression and weight changes in the first 12 months postpartum. Clin Endocrinol (Oxf). 2016 Dec;85(6):881-890. doi: 10.1111/cen.13150. Epub 2016 Aug 11. PMID 27374760
- [Background] Orta OR, Gelaye B, Bain PA, Williams MA. The association between maternal cortisol and depression during pregnancy, a systematic review. Arch Womens Ment Health. 2018 Feb;21(1):43-53. doi: 10.1007/s00737-017-0777-y. Epub 2017 Sep 24. PMID 28942465
- [Background] Wolfram M, Bellingrath S, Kudielka BM. The cortisol awakening response (CAR) across the female menstrual cycle. Psychoneuroendocrinology. 2011 Jul;36(6):905-12. doi: 10.1016/j.psyneuen.2010.12.006. Epub 2011 Jan 14. PMID 21237574
- [Background] Hodgson NA, Granger DA. Collecting saliva and measuring salivary cortisol and alpha-amylase in frail community residing older adults via family caregivers. J Vis Exp. 2013 Dec 18;(82):e50815. doi: 10.3791/50815. PMID 24378361
- [Background] Foody C, James JE, Leader G. Parenting stress, salivary biomarkers, and ambulatory blood pressure: a comparison between mothers and fathers of children with autism spectrum disorders. J Autism Dev Disord. 2015 Apr;45(4):1084-95. doi: 10.1007/s10803-014-2263-y. PMID 25287900
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Berry JO, Jones WH. The parental stress scale: Initial psychometric evidence. Journal of Social and Personal Relationships 1995;12:463-72
- [Background] Bourke-Taylor H, Law M, Howie L, Pallant JF. Development of the Child's Challenging Behaviour Scale (CCBS) for mothers of school-aged children with disabilities. Child Care Health Dev. 2010 Jul;36(4):491-8. doi: 10.1111/j.1365-2214.2009.01055.x. Epub 2009 Dec 29. PMID 20047597
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Crandal R. The measurement of self-esteem and related constructs, Pp. 80-82 in JP Robinson and PR Shaver (Eds), Measures of social psychological attitudes. Revised edition. Ann Arbor: ISR 1973.
- [Background] Gosling SD, Rentfrow PJ, Swann WB. A very brief measure of the Big-Five personality domains. Journal of Research in personality 2003;37:504-28.
- [Background] Hoffman L, Marquis J, Poston D, Summers JA, Turnbull A. Assessing Family Outcomes: Psychometric Evaluation of the Beach Center Family Quality of Life Scale. Journal of Marriage and Family 2006;68:1069-83.
- [Background] Lupien SJ, Seguin F. How to measure stress in humans. Centre for Studies in Human Stress 2013.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lyubomirsky S, Lepper HS. A measure of subjective happiness: Preliminary reliability and construct validation. Social indicators research 1999;46:137-55.
- [Background] Mak WWS, Cheung RYM. Affiliate Stigma Among Caregivers of People with Intellectual Disability or Mental Illness. J Appl Res Intellect Disabil 2008;21:532-45.
- [Background] Poston D, Turnbull A, Park J, Mannan H, Marquis J, Wang M. Family quality of life: a qualitative inquiry. Ment Retard. 2003 Oct;41(5):313-28. doi: 10.1352/0047-6765(2003)412.0.CO;2. PMID 12962536
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Tolan PH, Gorman-Smith D, Huesmann LR, Zelli A. Assessment of family relationship characteristics: A measure to explain risk for antisocial behavior and depression among urban youth. Psychological Assessment 1997;9:212.
- [Background] Yaneva M, Mosnier-Pudar H, Dugue MA, Grabar S, Fulla Y, Bertagna X. Midnight salivary cortisol for the initial diagnosis of Cushing's syndrome of various causes. J Clin Endocrinol Metab. 2004 Jul;89(7):3345-51. doi: 10.1210/jc.2003-031790. PMID 15240613
- [Background] El-Farhan N, Rees DA, Evans C. Measuring cortisol in serum, urine and saliva - are our assays good enough? Ann Clin Biochem. 2017 May;54(3):308-322. doi: 10.1177/0004563216687335. Epub 2017 Mar 16. PMID 28068807
- [Background] Kirschbaum C, Hellhammer DH. Salivary cortisol in psychoneuroendocrine research: recent developments and applications. Psychoneuroendocrinology. 1994;19(4):313-33. doi: 10.1016/0306-4530(94)90013-2. PMID 8047637
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Sammito S, Bockelmann I. Reference values for time- and frequency-domain heart rate variability measures. Heart Rhythm. 2016 Jun;13(6):1309-16. doi: 10.1016/j.hrthm.2016.02.006. Epub 2016 Feb 12. PMID 26883166
- [Background] Nunan D, Sandercock GR, Brodie DA. A quantitative systematic review of normal values for short-term heart rate variability in healthy adults. Pacing Clin Electrophysiol. 2010 Nov;33(11):1407-17. doi: 10.1111/j.1540-8159.2010.02841.x. PMID 20663071
- [Background] Giles D, Draper N, Neil W. Validity of the Polar V800 heart rate monitor to measure RR intervals at rest. Eur J Appl Physiol. 2016 Mar;116(3):563-71. doi: 10.1007/s00421-015-3303-9. Epub 2015 Dec 26. PMID 26708360
- [Background] Tarvainen MP, Niskanen JP, Lipponen JA, Ranta-Aho PO, Karjalainen PA. Kubios HRV--heart rate variability analysis software. Comput Methods Programs Biomed. 2014;113(1):210-20. doi: 10.1016/j.cmpb.2013.07.024. Epub 2013 Aug 6. PMID 24054542
- [Background] Urfer-Maurer N, Ludyga S, Stalder T, Brand S, Holsboer-Trachsler E, Gerber M, Grob A, Weber P, Lemola S. Heart rate variability and salivary cortisol in very preterm children during school age. Psychoneuroendocrinology. 2018 Jan;87:27-34. doi: 10.1016/j.psyneuen.2017.10.004. Epub 2017 Oct 5. PMID 29035709
- [Background] Hofmann B, Jacobs K, Navarrete Santos A, Wienke A, Silber RE, Simm A. Relationship between cardiac tissue glycation and skin autofluorescence in patients with coronary artery disease. Diabetes Metab. 2015 Nov;41(5):410-5. doi: 10.1016/j.diabet.2014.12.001. Epub 2014 Dec 29. PMID 25553578
- [Background] de Vos LC, Lefrandt JD, Dullaart RP, Zeebregts CJ, Smit AJ. Advanced glycation end products: An emerging biomarker for adverse outcome in patients with peripheral artery disease. Atherosclerosis. 2016 Nov;254:291-299. doi: 10.1016/j.atherosclerosis.2016.10.012. Epub 2016 Oct 6. PMID 27751506
- [Background] Grover-Paez F, Cardona-Munoz EG, Cardona-Muller D, Guzman-Saldivar VH, Rodriguez-De la Cerda M, Jimenez-Cazarez MB, Totsuka-Sutto SE, Alanis-Sanchez GA, Ramos-Becerra CG. Validation of the Omron HEM-7320-LA, upper arm blood pressure monitor with Intelli Wrap Technology Cuff HEM-FL1 for self-measurement and clinic use according to the European Society of Hypertension International Protocol revision 2010 in the Mexican population. Blood Press Monit. 2017 Dec;22(6):375-378. doi: 10.1097/MBP.0000000000000290. PMID 28945665
- [Background] Verberk WJ, Kessels AG, Thien T. Blood pressure measurement method and inter-arm differences: a meta-analysis. Am J Hypertens. 2011 Nov;24(11):1201-8. doi: 10.1038/ajh.2011.125. Epub 2011 Jul 21. PMID 21776035
- [Background] Ali BA, Abdelhakm AA, Abdelhameed MA, Tawfik NK. Quality of Life in Children with Type I Diabetes Mellitus (T1D) in Minia Governorate: Relationship with Mood and Family Attitudes. J Diabetes Metab 2017;8:5.
- [Background] Andrade EM, Geha LM, Duran P, Suwwan R, Machado F, do Rosario MC. Quality of Life in Caregivers of ADHD Children and Diabetes Patients. Front Psychiatry. 2016 Jul 25;7:127. doi: 10.3389/fpsyt.2016.00127. eCollection 2016. PMID 27504099
- [Background] Dardas LA, Ahmad MM. Quality of life among parents of children with autistic disorder: a sample from the Arab world. Res Dev Disabil. 2014 Feb;35(2):278-87. doi: 10.1016/j.ridd.2013.10.029. Epub 2013 Dec 4. PMID 24316492
- [Background] Gagliano A, Lamberti M, Siracusano R, Ciuffo M, Boncoddo M, Maggio R, Rosina S, Cedro C, Germano E. A Comparison between Children with ADHD and Children with Epilepsy in Self-Esteem and Parental Stress Level. Clin Pract Epidemiol Ment Health. 2014 Dec 24;10:176-83. doi: 10.2174/1745017901410010176. eCollection 2014. PMID 25614755
- [Background] Hullmann SE, Wolfe-Christensen C, Ryan JL, Fedele DA, Rambo PL, Chaney JM, Mullins LL. Parental overprotection, perceived child vulnerability, and parenting stress: a cross-illness comparison. J Clin Psychol Med Settings. 2010 Dec;17(4):357-65. doi: 10.1007/s10880-010-9213-4. PMID 21086027
- [Background] Leung C, Tsang SK. The Chinese Parental Stress Scale: psychometric evidence using Rasch modeling on clinical and nonclinical samples. J Pers Assess. 2010 Jan;92(1):26-34. doi: 10.1080/00223890903379209. PMID 20013453
- [Background] Manee F, Ateya Y, Rassafiani M. A Comparison of the Quality of Life of Arab Mothers of Children with and without Chronic Disabilities. Phys Occup Ther Pediatr. 2016 Aug;36(3):260-71. doi: 10.3109/01942638.2015.1076558. Epub 2015 Nov 13. PMID 26566139
- [Background] Mugno D, Ruta L, D'Arrigo VG, Mazzone L. Impairment of quality of life in parents of children and adolescents with pervasive developmental disorder. Health Qual Life Outcomes. 2007 Apr 27;5:22. doi: 10.1186/1477-7525-5-22. PMID 17466072
- [Background] Norizan A, Shamsuddin K. Predictors of parenting stress among Malaysian mothers of children with Down syndrome. J Intellect Disabil Res. 2010 Nov;54(11):992-1003. doi: 10.1111/j.1365-2788.2010.01324.x. Epub 2010 Sep 27. PMID 20868445
- [Background] Phillips BA, Conners F, Curtner-Smith ME. Parenting children with down syndrome: An analysis of parenting styles, parenting dimensions, and parental stress. Res Dev Disabil. 2017 Sep;68:9-19. doi: 10.1016/j.ridd.2017.06.010. Epub 2017 Jul 7. PMID 28692948
- [Background] Roncada C, Dias CP, Goecks S, Cidade SE, Pitrez PM. [Usefulness of the WHOQOL-BREF questionnaire in assessing the quality of life of parents of children with asthma]. Rev Paul Pediatr. 2015 Jul-Sep;33(3):268-74. doi: 10.1016/j.rpped.2015.01.007. Epub 2015 Jun 9. PMID 26137868
- [Background] Semakina NV, Mikhailov VA, Bagaev VI. Assessing the quality of life of families of children with epilepsy. Obozrenie psikhiatrii i meditsinskoi psikhologii im VM Bekhtereva 2012:73-6.
- [Background] Vadakedom SS, Antony JM, Padma BK, Mammen DS, Thankappan BP. Quality of life of mothers of children with Down syndrome. J Evol Med Dent Sci-JEMDS 2017;6:2939-42.
- [Background] Wolf JM, Miller GE, Chen E. Parent psychological states predict changes in inflammatory markers in children with asthma and healthy children. Brain Behav Immun. 2008 May;22(4):433-41. doi: 10.1016/j.bbi.2007.10.016. Epub 2007 Dec 18. PMID 18068332
- [Background] Epifanio MS, Genna V, Vitello MG, Roccella M, La Grutta S. Parenting stress and impact of illness in parents of children with coeliac disease. Pediatr Rep. 2013 Dec 19;5(4):e19. doi: 10.4081/pr.2013.e19. eCollection 2013. PMID 24416498
- [Background] Scheier MF, Carver CS, Bridges MW. Distinguishing optimism from neuroticism (and trait anxiety, self-mastery, and self-esteem): a reevaluation of the Life Orientation Test. J Pers Soc Psychol. 1994 Dec;67(6):1063-78. doi: 10.1037//0022-3514.67.6.1063. PMID 7815302
- [Background] Monteagudo C, Mariscal-Arcas M, Rivas A, Lorenzo-Tovar ML, Tur JA, Olea-Serrano F. Proposal of a Mediterranean Diet Serving Score. PLoS One. 2015 Jun 2;10(6):e0128594. doi: 10.1371/journal.pone.0128594. eCollection 2015. PMID 26035442
- [Background] Bassett DR Jr. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1396. doi: 10.1249/01.MSS.0000078923.96621.1D. No abstract available. PMID 12900695
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Chung F, Subramanyam R, Liao P, Sasaki E, Shapiro C, Sun Y. High STOP-Bang score indicates a high probability of obstructive sleep apnoea. Br J Anaesth. 2012 May;108(5):768-75. doi: 10.1093/bja/aes022. Epub 2012 Mar 8. PMID 22401881
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Stelmach-Mardas M, Iqbal K, Mardas M, Kostrzewska M, Piorunek T. Clinical Utility of Berlin Questionnaire in Comparison to Polysomnography in Patients with Obstructive Sleep Apnea. Adv Exp Med Biol. 2017;980:51-57. doi: 10.1007/5584_2017_7. PMID 28255917